CLINICAL TRIAL: NCT04028141
Title: Prospective Observational Evaluation of a New Protocol for Adult Procedural Sedation With Ketamine-propofol in a 1 on 4 Ratio at the Emergency Department of a Tertiary Hospital
Brief Title: Evaluation of a New Protocol for Adult Procedural Sedation With Ketamine-propofol in a 1 on 4 Ratio
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201834755
Record Dates: First submitted 2019-06-05; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Procedural Sedation and Analgesia
Keywords: ketofol; propofol; ketamine; emergency department
MeSH Terms: conditions — Agnosia; Emergencies | interventions — Propofol; Ketamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- participants undergoing procedural sedation: The study gathered observational data about participants who underwent procedural sedation according to the new standard protocol with ketofol in a 1 on 4 concentration.
  The participant was observed for complications or cardiorespiratory interventions by the sedating physician until he was fully awake. Thirty minutes after the awakening, the participant was questioned for his remembrance and perception of the sedation and procedure. He was observed for complications until discharge
  Interventions: Drug: Procedural sedation with ketofol in a 1 on 4 ratio

INTERVENTIONS:
Drug: Procedural sedation with ketofol in a 1 on 4 ratio — The participant was brought to a zone where advanced life support could be optimally administered and where all necessary drugs and materials for treatment of complications are present. Oxygen saturation, continuous electrocardiogram, intermittent blood pressure measurement (every 2 minutes) and capnography were applied. A 20 gauge intravenous line was inserted. The participant was placed in semi-recumbent position and was given oxygen for at least 3 minutes through a non-rebreather mask unless contra-indications applied.
  Ketofol 1 on 4 was prepared by mixing 1ml of ketamine (50mg) and 20ml of propofol (200mg) in a single syringe. It was administrated as a loading dose of 1ml/10kg, corresponding to 0,952mg/kg propofol and 0,238mg/kg ketamine, and followed by titration in aliquots of 0,5ml/10kg every 1 to 2 minutes until desired depth of sedation was achieved, and then every 3-5 minutes to retain the desired depth of sedation. The loading dose was halved if above 65 years.
  Other Names: Propofol; Ketamine; Ketofol

SUMMARY:
Procedural sedation is the monitored use of sedatives and/or analgesics in a patient who must endure a short painful or frightening procedure, bringing the patient into a sedative state while retaining his spontaneous breathing and respiratory reflexes. Examples of these procedures are cardioversion, repositioning of a shoulder luxation or incision of a skin abscess, and these are frequently performed at the emergency ward. An easy and unambiguous protocol for procedural sedation was composed at the emergency department of the University Hospital of Ghent applicable for nearly all patients and procedures. This protocol included recommendations for necessary monitoring such as continuous electrocardiogram, intermittent blood pressure measurements, oxygen saturation and capnography, as well as safety precautions for standby medications or medical devices for hemodynamic and airway control. As sedative drug a mixture of ketamine and propofol ("ketofol") in a 1 on 4 ratio was selected based on the available literature. Both ketamine and propofol are known to neutralise each other's undesirable effects and ketamine adds an analgesic quality. Ketofol has proven effective and safe in studies and is non-inferior to propofol. Though it is most often used in a 1 on 1 ratio, both pharmacological and clinical studies favour a 1 on 4 ratio.

An adult patient presenting at the investigating hospital in need of procedural sedation, who agreed the informed consent for procedural sedation was treated according to this protocol. Patients with an American Society of Anesthesiologist physical status classification system status of III or more, with an anticipated difficult airway or intoxicated patients were discussed with the anaesthesiology department to decide the feasibility of sedation in the emergency ward setting. Pregnant patients were excluded.

Associated to this newly implemented protocol, an observational prospective study was associated to verify the safety and effectivity, and to score the physicians satisfaction. A separate informed consent was obtained for participation in the study to permit inclusion of patient and procedural data into a registry. Data was registered by the physician responsible for the sedation in a questionnaire. The investigators hypothesized the protocol with ketofol in a 1 on 4 ratio would be safe and effective and would serve to facilitate procedural sedation by emergency physicians.

DETAILED DESCRIPTION:
Procedural sedation is the monitored use of sedatives and/or analgesics in a patient who must endure a short painful or frightening procedure, bringing the patient into a sedative state while retaining his spontaneous breathing and respiratory reflexes. Examples of these procedures are cardioversion, repositioning of a shoulder luxation or incision of a skin abscess, and these are frequently performed at the emergency ward. An easy and unambiguous protocol for procedural sedation was composed at the emergency department of the University Hospital of Ghent applicable for nearly all patients and procedures. This protocol included recommendations for necessary monitoring such as continuous electrocardiogram, intermittent blood pressure measurements, oxygen saturation and capnography, as well as safety precautions for standby medications or medical devices for hemodynamic and airway control. As sedative drug a mixture of ketamine and propofol ("ketofol") in a 1 on 4 ratio was selected based on the available literature. Both ketamine and propofol are known to neutralise each other's undesirable effects and ketamine adds an analgesic quality. Ketofol has proven effective and safe in studies and is non-inferior to propofol. Though it is most often used in a 1 on 1 ratio, both pharmacological and clinical studies favour a 1 on 4 ratio. According to the protocol ketofol 1 on 4 was prepared by mixing 1ml of ketamine (50mg) and 20ml of propofol (200mg) in a single syringe and administrated as a loading dose of 1ml/10kg, followed by a stepwise titration in aliquots of 0,5ml/10kg. Above 65 years the loading dose was halved.

An adult patient presenting at the investigating hospital in need of procedural sedation, who agreed the informed consent for procedural sedation was treated according to this protocol. Patients with an American Society of Anesthesiologist physical status classification system status of III or more, with an anticipated difficult airway or intoxicated patients were discussed with the anaesthesiology department to decide the feasibility of sedation in the emergency ward setting. Pregnant patients were excluded.

Associated to this newly implemented protocol, an observational prospective study was associated to verify the safety and effectivity, and to score the physicians satisfaction. A separate informed consent was obtained for participation in the study to permit inclusion of patient and procedural data into a registry. Data was registered by the physician responsible for the sedation in a questionnaire. The investigators hypothesized the protocol with ketofol in a 1 on 4 ratio would be safe and effective and would serve to facilitate procedural sedation by emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients presenting to the university hospital of Ghent and in need of procedural sedation as determined by the treating physician, who underwent procedural sedation by the standard protocol using ketofol in a 1 on 4 ratio.

Exclusion Criteria:

* pregnant patient
* procedural sedation not performed at the emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department of the University Hospital of Ghent, a tertiary hospital with over 1000 acute beds.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Respiratory complication or intervention | From start of sedation, until half an hour after participant woke up from sedation ( participant fully communicative and obedient for commands). On average a total monitoring time of 40 minutes.
  * Complication: desaturation (< 92%), apnea (absent end-tidal CO2 for > 15s and no breathing movements), hypoventilation (respiratory frequency < 8 /minute), airway obstruction (absent end-tidal CO2 for > 15s and breathing movements), laryngospasm (partial or complete airway obstruction, not responding to airway repositioning or introduction of naso- or oropharyngeal cannula), aspiration due to vomiting
  * Intervention: airway repositioning (head tilt or chin lift), pain stimulus for breathing stimulation, introduction of naso- or oropharyngeal cannula, positive pressure ventilation, introduction of laryngeal mask or endotracheal tube
Hemodynamic complication or intervention | From start of sedation, until half an hour after participant woke up from sedation ( participant fully communicative and obedient for commands). On average a total monitoring time of 40 minutes.
  * Complication: hypotension (systolic blood pressure less than 90mmHg, or drop of 10% of systolic blood pressure )
  * Intervention: fluid bolus given, use of inotropes

SECONDARY OUTCOMES:
Success of procedure | From start of sedation, until participant woke up from sedation ( participant fully communicative and obedient for commands). Assessment was made at time of awakening
  sedation adequate for performing procedure (yes/no)
Amnesia | Assessed 30 minutes after awakening ( participant fully communicative and obedient for commands) and addressing the moment of performance of the procedure during sedated state
  amnesia of the procedure by the patient (yes/no)
Agitation or hallucination | From start of sedation, until half an hour after participant woke up from sedation ( participant fully communicative and obedient for commands). On average a total monitoring time of 40 minutes.
  * Agitation during or after sedation (yes/no)
  * Hallucination during or after sedation (yes/no)
    * If hallucination: Pleasant / neutral / unpleasant
Duration of sedation | Start of sedation until awakening ( participant fully communicative and obedient for commands)
  Time from start of sedation till completely awake, expressed in minutes
Satisfaction sedating physician | Assessed 30 minutes after awakening ( participant fully communicative and obedient for commands), concerning the period from start of sedation until 30 minutes after awakening
  - satisfaction of the sedation with the current protocol, score on a five point Likert scale (++ / + / + - / - / - - , meaning very satisfied / satisfied / neither satisfied nor dissatisfied / dissatisfied / very dissatisfied )

OTHER OUTCOMES:
American Society of Anesthesiologist physical status classification status participant | start of procedure
  American Society of Anesthesiologist physical status classification status I, II, III of IV
Age of participant | start of procedure
  Age of participant in years
Type of procedure | start of procedure
  * Reduction of luxation or fracture ( shoulder, ankle/foot, hip, elbow, other … (possibility to fill in))
  * Abscess incision
  * Cardioversion
  * Chest drain placement
  * Other: … (possibility to fill in)

CONTACTS AND LOCATIONS:
Overall Officials: Peter De Paepe, PhD, MD, Principal Investigator — University Hospital of Ghent
Locations (1):
- University Hospital of Ghent - Emergency Department, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No
Informed consent included statement of anonymity and no standard public access to data collected.

REFERENCES:
- [Background] Miner JR, Moore JC, Austad EJ, Plummer D, Hubbard L, Gray RO. Randomized, double-blinded, clinical trial of propofol, 1:1 propofol/ketamine, and 4:1 propofol/ketamine for deep procedural sedation in the emergency department. Ann Emerg Med. 2015 May;65(5):479-488.e2. doi: 10.1016/j.annemergmed.2014.08.046. Epub 2014 Oct 16. PMID 25441247
- [Background] Ferguson I, Bell A, Treston G, New L, Ding M, Holdgate A. Propofol or Ketofol for Procedural Sedation and Analgesia in Emergency Medicine-The POKER Study: A Randomized Double-Blind Clinical Trial. Ann Emerg Med. 2016 Nov;68(5):574-582.e1. doi: 10.1016/j.annemergmed.2016.05.024. Epub 2016 Jul 22. PMID 27460905
- [Background] Yan JW, McLeod SL, Iansavitchene A. Ketamine-Propofol Versus Propofol Alone for Procedural Sedation in the Emergency Department: A Systematic Review and Meta-analysis. Acad Emerg Med. 2015 Sep;22(9):1003-13. doi: 10.1111/acem.12737. Epub 2015 Aug 20. PMID 26292077
- [Background] Jalili M, Bahreini M, Doosti-Irani A, Masoomi R, Arbab M, Mirfazaelian H. Ketamine-propofol combination (ketofol) vs propofol for procedural sedation and analgesia: systematic review and meta-analysis. Am J Emerg Med. 2016 Mar;34(3):558-69. doi: 10.1016/j.ajem.2015.12.074. Epub 2015 Dec 29. PMID 26809929
- [Background] Andolfatto G, Abu-Laban RB, Zed PJ, Staniforth SM, Stackhouse S, Moadebi S, Willman E. Ketamine-propofol combination (ketofol) versus propofol alone for emergency department procedural sedation and analgesia: a randomized double-blind trial. Ann Emerg Med. 2012 Jun;59(6):504-12.e1-2. doi: 10.1016/j.annemergmed.2012.01.017. Epub 2012 Mar 7. PMID 22401952
- [Background] Godwin SA, Caro DA, Wolf SJ, Jagoda AS, Charles R, Marett BE, Moore J; American College of Emergency Physicians. Clinical policy: procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2005 Feb;45(2):177-96. doi: 10.1016/j.annemergmed.2004.11.002. No abstract available. PMID 15671976

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT04028141/Prot_SAP_ICF_000.pdf